CLINICAL TRIAL: NCT04189887
Title: Effect of a Single Bout of Aerobic Exercise on Implicit Sequence Learning in People With Parkinson's Disease
Brief Title: Single Bout Exercise on Learning in PD
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20190901RINC
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PD+AEX: The group of people with PD which will perform aerobic exercise after motor skill acquisition
  Interventions: Behavioral: aerobic exercise (cycling); Behavioral: Implicit sequence learning
- PD-AEX: The group of people with PD which will not perform aerobic exercise after motor skill acquisition
  Interventions: Behavioral: Implicit sequence learning
- CON+AEX: The group of control participants which will perform aerobic exercise after motor skill acquisition
  Interventions: Behavioral: aerobic exercise (cycling); Behavioral: Implicit sequence learning
- CON-AEX: The group of control participants which will not perform aerobic exercise after motor skill acquisition
  Interventions: Behavioral: Implicit sequence learning

INTERVENTIONS:
Behavioral: aerobic exercise (cycling) — People who perform aerobic exercise will ride on a stationary bike for 20 minutes after motor skill learning
  Groups: CON+AEX; PD+AEX
Behavioral: Implicit sequence learning — All participants will practice the serial reaction time task (SRTT) on the first day, and retention performance will be assessed immediately, on the 2nd day, and on the 7th day of study.
  Other Names: serial reaction time task (SRTT)

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder associated with a loss of dopamine in the basal ganglia and is characterized by several cardinal motor signs. In addition to the commonly recognized motor symptoms, cognitive impairments are also often observed in people with PD. Unlike motor deficits, cognitive impairments are not always responsive to dopaminergic treatment. While medication may ameliorate some cognitive dysfunctions (e.g., executive function), it may exacerbate others (e.g., motor learning). Therefore, it is crucial for clinicians to look for treatment approaches, other than medication, to enhance cognitive function. In this proposed study, the investigators are especially interested in determining a method to enhance motor learning ability in people with PD.

Motor learning deficits in people with PD have been well established through different tasks including motor adaptation task such as maintain balance on a stabilometer or motor sequence task such as performing a serial reaction time task (SRTT). Motor sequence learning is important in acquiring real-life motor skill such as tying shoes laces. Based on the past evidences, people with PD have impairments in motor sequence learning, particularly in implicit sequence learning. Since implicit motor sequence learning constitutes a critical part of everyday activities such as typing and changing clothes, establishing an approach to enhance implicit sequence learning is important.

In the literature conducted with non-disable adults, one of the most effective method to enhance motor learning is aerobic exercise. Only one study, to the best of knowledge, has investigated the effect of aerobic exercise on learning to maintain balance on a stabilometer in people with PD. To date, no study has investigated whether a single bout of aerobic exercise could improve implicit sequence learning in PD. Therefore, the goal of this proposed study is to investigate the effect of a single bout of aerobic exercise on implicit sequence learning and the associated neurophysiological changes in people with PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a neurodegenerative disorder associated with loss of dopamine in the basal ganglia and is characterized by several cardinal motor signs, such as tremor, rigidity, bradykinesia, and postural instability. In addition to the commonly recognized motor symptoms, non-motor symptoms such as olfactory dysfunction, emotional issues, autonomic dysfunction and cognitive impairments are also often observed in people with PD. Among these non-motor symptoms, cognitive dysfunction is the most disturbing deficit and can hugely affect an individual's daily activity. Unlike motor deficits, these cognitive impairments are not always responsive to dopaminergic treatment. While medication may ameliorate some cognitive dysfunctions (e.g., executive function), it may exacerbate others (e.g., motor learning).Therefore, it is crucial for clinicians to look for treatment approaches, other than medication, to enhance cognitive function . In this proposed study, the investigators are especially interested in determining a method to enhance motor learning ability and reduce motor learning deficit in people with PD as motor learning is a crucial basis in learning new skills and optimizing activities of daily living.

Motor learning deficits in people with PD have been well established through different tasks including motor adaptation task such as maintain balance on a stabilometer or motor sequence task such as performing a serial reaction time task (SRTT). Motor sequence learning is important in acquiring real-life motor skill such as tying shoes laces and using chopsticks. There are two types of experiment paradigms to assess motor sequence learning, they are implicit sequence task and explicit sequence task. Compared with age-matched non-disable adults, people with PD demonstrated different level of impairments in learning those tasks. In this study, the investigators will especially focus on the impairment in motor sequence learning in people with PD. Based on the evidences, implicit sequence learning is more affected in people in PD compared to explicit sequence learning. Since implicit motor sequence learning constitutes a critical part of everyday activities such as typing and changing clothes, therefore the investigators are more interested in exploring implicit sequence learning in people with PD.

As previously reviewed, motor learning dysfunction could not be ameliorated by dopaminergic intake, thus several researchers aimed to find alternative method to improve motor learning ability. In the literature conducted with non-disable adults, one of the most effective method to enhance motor learning is aerobic exercise.7 Rhee et al. (2016) conducted a study and showed that a single bout of 20 minutes high intensity aerobic exercise can improve the performance of a finger sequence learning task in non-disable adults. Only one study, to the best of our knowledge, has investigated the effect of aerobic exercise on learning to maintain balance on a stabilometer in people with PD. The participants with PD were required to perform a single bout of 30-minute moderate intensity (60-70% VO2max) cycling exercise before practicing the stabilometer task. Their results found that compared to the non-aerobic condition, 30 minutes of aerobic exercise led to great improvements in motor performance at retention. However, there are some limitations of this study which may influence the result. First of all, 30 minutes of aerobic exercise before skill learning might be too fatiguing for people with PD, and might compromise subsequent practice of the stabilometer task. Furthermore, the authors found improvements in maintaining balance on a stabilometer but the related neurophysiological changes have not been determined. Therefore, the goal of this proposed study is to modify the above limitations and to conduct a study to investigate the effect of a single bout of aerobic exercise to implicit sequence learning and the related neurophysiological changes in people with PD. More importantly, the investigatorse would like to investigate whether corticomotor excitability will change along with motor learning improvement in people with PD.

The purpose of this proposed study is to explore whether a single-bout aerobic exercise could enhance implicit motor sequence learning in people with PD. Moreover, the neurophysiological changes associated with aerobic exercise and learning will be determined.

ELIGIBILITY:
Inclusion Criteria:

* 1) able to follow instructions to perform the tasks
* 2) without other neurological disorders in addition to PD
* 3) no surgery or injury of the upper extremities in recent 6 months

Exclusion Criteria:

* 1) deep brain stimulation or pacemaker implanted
* 2) a self-history of seizure
* 3) unstable medical conditions
* 4) a blood-relative with a history of epilepsy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed of idiopathic PD and non-disabled age-matched controls will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-09-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Performance of the sequence learning task | 30 minutes
  A serial reaction time task (SRTT) will be used to determine the sequence learning ability. At the beginning of the SRTT, only one circle will be filled with color while others remain hollow. Once the participants hit the correct button, the next target will appear. Unknown to the participants, an 12-element sequence is embedded within the random sequences. The response time of the key presses of the embedded sequence will be recorded. The change score will be calculated between the 1st and 2nd sessions, and between the 1st and 7th sessions.

SECONDARY OUTCOMES:
Corticomotor excitability | 50 minutes
  Transcranial magnetic stimulation (TMS) will be used to evaluate corticomotor excitability. Corticomotor excitability outcomes will include motor evoke potential (MEP), cortical silent period (CSP) duration, short-interval intracortical inhibition (SICI), intracortical facilitation (ICF), and long-interval intracortical inhibition (LICI). The RMT could reflect the membrane excitability of the corticospinal neurons and the cortical interneurons. Peak-to-peak MEP amplitude is an indicator of the integrity and excitability of the corticospinal tract. The CSP is a period when EMG activity being suppressed for a few hundred milliseconds after the MEP, and has often been used as an indicator of the inhibitory mechanism occurs within the corticospinal tract. The SICI, ICF, and LICI have been identified to be good indicators of intracortical inhibition and facilitation.

OTHER OUTCOMES:
Montreal Cognitive Assessment | 10 minutes
  Montreal Cognitive Assessment (MoCA) will be to used to assess general cognitive function of the participants. The total score of MoCA ranges from 0 to 30 and a higher score suggests better cognitive function. The MoCA has good to excellent psychometric properties (sensitivity 90% and specificity 75%), and has been proven as a suitable and accurate standard for screening all levels of cognition for individuals with PD.
Stroop test | 5 minutes
  Stroop test will be used to assess the ability to inhibit cognitive interference. The participants will be instructed to read out the ink color of the word, but not the color word name, as accurately and as fast as possible within 45 seconds. The more the participants read out correctly, the better they are.
The Trail Making test | 5 minutes
  The Trail Making Test will be used to assess the ability of visual attention and task switching. Participants will be required to connect alternatively between the numbers and the letters (e.g., 1-rat-2-ox-3-tiger …, etc.) as accurately and as fast as possible. The time taken to finish the test will be recorded and the shorter time suggests better performance.
The Unified Parkinson's Disease Rating Scale | 15 minutes
  Only the part 3 of the The Unified Parkinson's Disease Rating Scale (UPDRS) will be assessed. It is focus on the motor function. The total score of part 3 ranges from 0 to 72.The higher the score, the more severe the patient is.
The New Freezing of Gait Questionnaire | 5 minutes
  The New Freezing of Gait Questionnaire (NFOG-Q) will be used to evaluate the freezing frequency and severity of the patients with PD. The total score of NFOG-Q ranges from 0-28.The higher the score, the more severe freezing of gait the patient is suffering from.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Yun Lee, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongcheng, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan ST, Tai CH, Wang LY, Luh JJ, Lee YY. Influences of Aerobic Exercise on Motor Sequence Learning and Corticomotor Excitability in People With Parkinson's Disease. Neurorehabil Neural Repair. 2023 Jan;37(1):37-45. doi: 10.1177/15459683221147006. Epub 2023 Jan 12. PMID 36636767